CLINICAL TRIAL: NCT06536946
Title: Expression of B-catenin in Cutaneous Squamous Cell Carcinoma and Its Mimickers
Brief Title: B-catenin in Cutaneous Squamous Cell Carcinoma and Its Mimickers
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nermin Sarwat Habib, Teaching assistant of pathology, Sohag University
Other Study IDs: Soh-Med-25-05-07MS
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: B-catenin; Cutaneous squamous cell carcinoma; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 50 formalin fixed parrafin embedded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: 50 formalin fixed parrafin embedded tissue blocks of cutaneous squamous cell carcinoma and its mimickers , from each block 2 tissue section; one tissue section stained by Hematoxilin and Eoisin and other tissue section will be stained immunohistochemically by anti human B-catenin
  Interventions: Biological: Immunohistochemical staining

INTERVENTIONS:
Biological: Immunohistochemical staining — Staining of cutanous squamous cell carcinoma and its mimickers by monoclonal antibodies against human B-catenin by immunohistochemical procedures

SUMMARY:
Examine the role of B-catenin in differentiation of cutaneous squamous cell carcinoma from other lesions that may be similar to it

DETAILED DESCRIPTION:
Skin cancer is one of the most common form of cancer worldwide. Cutaneous squamous cell carcinoma is one of most common skin tumers that caused by many factors as ultra violet ,ionizing radiation and others . It was an advanced spectrum ranging from actinic keratosis to invasive and metastatic squmous cell carcinoma. Correct identification of cutaneous squamous cell carcinoma is a challenge as it has both clinically and histopathologically mimickers.

So the aim of this study is to identify the expression of B-catenin in cutaneous Squamous cell carcinoma and its mimickers.

ELIGIBILITY:
Inclusion Criteria:

* tissue blocks with sufficient materials Cases with sufficient data

Exclusion Criteria:

* tissue blocks with insufficient and necrotic materials. Casas with insufficient data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: archived formalin fixed parrafin embedded tissue pieces of patients of cutanous squamous cell carcinoma and its mimickers admitted to sohag University hospital from period juniory 2023 to June 2024
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Detection of B-catenin expression in cutanous squamous cell carcinoma and its mimickers | 6 month
  Detection of expression of B-catenin in cutaneous squamous cell carcinoma and its mimickers by immunohistochemical procedures using antihuman B-catenin monoclonal antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided